CLINICAL TRIAL: NCT01973192
Title: Viral Pathogenesis of Early Cystic Fibrosis Lung Disease
Acronym: Early CF
Status: Completed | Type: Observational
Sponsor: Indiana University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Stephanie D. Davis, MD, Section Director of Pediatric Pulmonology, Allergy and Sleep Medicine, Indiana University
Organization: Indiana University (Other)
Other Study IDs: 1R01HL116211-01 (NIH); 1R01HL116211-01 (NIH)
Record Dates: First submitted 2013-09-17; First posted 2013-10-31 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Urea, Bronchopulmonary Lavage samples, Nasal swabs and Oral swabs, Stool samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to test the hypothesis that early viral infections alter the bacterial flora and inflammatory profile in the airway and accelerate progression of pulmonary disease in infants with cystic fibrosis.

DETAILED DESCRIPTION:
The proposed study is a unique international collaboration between three large CF research centers. This proposal will determine the impact of early respiratory viral infections on bacterial flora and inflammatory profiles in the CF airway as well as the impact of these pathogens on clinical, physiologic and structural markers of disease.The proposed study is designed to follow infants diagnosed with CF through newborn screening to determine the effect of viral infections on the lower airway microbiome, clinical symptoms, pulmonary function and structural changes during the first year of life. The proposed study will measure lower airway inflammation and infection using BAL, oral swabs, and nasal swabs; outcomes will be assessed through infant lung function testing, computerized tomography scans of the chest, and pulmonary exacerbation rate.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of CF by newborn screening, at least one clinical feature of CF, and documented sweat chloride greater than 60 mEq/L by quantitative pilocarpine iontophoresis or compatible genotype with two identifiable mutant CFTR alleles.
2. Less than 4 months of age at Screening Visit
3. Ability to comply with study visits and study procedures as judged by site investigator.

Exclusion Criteria:

1. Intercurrent respiratory illness, defined as increase in cough, wheezing, or respiratory rate with onset 14 days before iPFT-bronchoscopy visit.
2. Measured hemoglobin oxygen saturation less than 95% during the iPFT-bronchoscopy visit.
3. History of adverse reaction to sedation.
4. Clinically significant upper airway obstruction as determined by the site investigator.
5. Severe gastroesophageal reflux, defined as persistent frequent emesis despite therapy.
6. Major organ dysfunction, not including pancreatic dysfunction.
7. Physical findings that would compromise the safety of the subject or the quality of the study data as determined by site investigator.

Ages: 2 Months to 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants, less than 4 months of age who have been diagnosed with Cystic Fibrosis
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2013-05; Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Viral infection | 12 months
  To determine the effect(s) of viral infections on the evolution of endobronchial bacterial infection and inflammation in CF infants.

SECONDARY OUTCOMES:
Pulmonary exacerbation rate | 12 Months
  To identify the impact of respiratory viruses on the onset, frequency, and duration of respiratory symptoms in CF infants diagnosed through newborn screening.
Forced Expiratory Volume | 12 months
  To assess development of early lung disease as defined through physiological measures of forced expiratory flows, lung volumes, and ventilation inhomogeneity in CF infants.

OTHER OUTCOMES:
Bronchiectasis | 12 Months
  To evaluate the association of early viruses on the development of early lung disease in CF infants as defined through comprehensive structural and airway modeling techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie D. Davis, MD, Principal Investigator — Indiana University School of Medicine
Locations (4):
- United States (2):
  - Riley Hospital for Children at Indiana University Health, Indianapolis, Indiana
  - St. Louis Children's Hospital, St Louis, Missouri
- Australia (2):
  - The Royal Children's Hospital, Melbourne, Victoria
  - Telethon Kids Institute, West Perth